CLINICAL TRIAL: NCT07247838
Title: Investigation Into the Gut Microbiota-Immune-Inflammatory Interaction Network and Its Mechanisms in Patients With Ischemic Stroke
Brief Title: Prospective Cohort Control Study on Changes in Gut Microbiota in Ischemic Stroke
Status: Recruiting | Type: Observational
Sponsor: Affiliated Hospital of Nantong University (Other)
Collaborators: Zhejiang University (Other)
Responsible Party: Principal Investigator, Yongtao Gao, Deputy Director of the Anesthesiology Department, Affiliated Hospital of Nantong University
Other Study IDs: 2025-k257-01
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Ischemic Stroke
Keywords: Gut Microbiota
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stroke group: 1. For patients with acute ischemic stroke for the first time, the time from symptom onset to hospitalization and completion of the first sample collection was within 48 hours;
  2. Over 18 years old, male or female;
  3. Patients with ischemic stroke who scored ≥4 on the National Institutes of Health Stroke Scale (NIHSS);
- Healthy Volunteer Group: Healthy volunteers with no history of ischemic stroke

SUMMARY:
1. Stroke stands as one of the leading causes of death and long-term disability worldwide, imposing a substantial socioeconomic burden. Annual new stroke cases are estimated between 9.5 million and 10.6 million. Stroke survivors commonly face challenges of poor long-term functional outcomes and compromised immunity, which not only drive quality-of-life deterioration but also fuel the persistent escalation of socioeconomic burdens. However, current clinical treatments for stroke prognosis improvement remain limited. In recent years, with the emergence of the "microbiota-gut-brain axis" concept and advancing research, the role of gut microbiota in stroke onset, progression, and prognosis regulation has garnered increasing attention.

   The gut-brain axis is a complex bidirectional communication network connecting the central nervous system with the gut and its microbiota, centered on the integration of the microbiota-gut-brain axis concept. Its signaling mechanisms primarily involve multiple pathways including neural (e.g., vagus nerve), endocrine (e.g., HPA axis and gut hormones), immune (e.g., cytokines), and microbial metabolic pathways (e.g., short-chain fatty acids (SCFAs) and neuroactive substances). Dysregulation of the gut-brain axis has been proven closely associated with various diseases, including irritable bowel syndrome (IBS) characterized by visceral hypersensitivity and motility abnormalities, inflammatory bowel disease (IBD) often accompanied by emotional comorbidities, autism spectrum disorder (ASD) with gastrointestinal symptoms and behavioral core symptoms, depression and anxiety related to microbiota dysbiosis and inflammation, as well as Parkinson's disease (PD) with pathological origins potentially originating in the gut. Recent studies support that gut microbiota interact with ischemic stroke through the gut-brain axis, thereby modulating stroke pathogenesis. Gut microbiota can regulate innate and adaptive immune responses and their derived metabolites through neural pathways, influencing host brain function and behavior. Gut microbiota metabolites-short-chain fatty acids (SCFAs) such as butyrate-reduce neuroinflammation and brain injury by promoting regulatory T cell differentiation and secretion of anti-inflammatory factors IL-10 and TGF-β, suppressing pro-inflammatory Th1/Th17 responses, and enhancing expression of blood-brain barrier tight junction proteins Occludin and ZO-1.

   Compared to traditional stroke treatments, gut microbiota therapy breaks the time window limitation. Even days after stroke, restoring a youthful gut microbiome can reduce neuroinflammation and promote recovery in stroke patients. This effect is largely mediated by metabolites produced by bacteria, particularly short-chain fatty acids.

   Although existing studies have demonstrated the crucial role of gut microbiota in stroke treatment, the mechanisms underlying its effects on improving physiological and behavioral functions in stroke patients, as well as the underlying mechanisms, remain insufficiently explored.
2. Purpose of this study To investigate the mechanisms by which gut microbiota and their metabolites improve the physiological and neurological functions of stroke patients, and to provide new therapeutic approaches for improving the prognosis of stroke patients.
3. Research Design 3.1 Research Methodology This is a single-center, non-interventional, cohort-controlled clinical study that randomly enrolled 100 stroke patients and 100 healthy individuals. The participants were divided into a stroke group (case group, CS group) and a healthy control group (CON group), with 100 cases in each group. The primary objectives were to investigate the gut microbiota composition, intestinal barrier function, and inflammatory cytokine levels in stroke patients versus healthy controls, while exploring the mechanisms of beneficial gut microbiota in stroke recovery. This research may provide new therapeutic approaches to address current treatment limitations.

DETAILED DESCRIPTION:
Recent advancements in stroke treatment have been remarkable, yet numerous challenges persist. The primary objective of acute ischemic stroke management remains early restoration of cerebral perfusion, achieved through thrombolysis (intravenous or mechanical), thrombectomy, or their combination, followed by transfer to specialized stroke units for comprehensive care. As the gold standard for acute ischemic stroke, rt-PA (alteplase) is the only thrombolytic approved by major global regulators. Despite over 25 years of clinical use, this therapy still faces limitations including a narrow therapeutic window (typically within 4.5 hours of onset), risks of symptomatic intracranial hemorrhage, ineffectiveness in infarcted tissue, individual response variability, and multiple contraindications. While rt-PA remains the most recognized treatment for acute ischemic stroke within 4.5 hours, its clinical cure rate is not 100%. Some patients not only fail to improve neurological deficits but experience aggravated symptoms, resulting in severe psychological distress, significant quality-of-life impairment, and substantial financial burdens for families. Although thrombectomy has extended the therapeutic window from 6 hours to 24 hours in some cases, the "time is brain" principle remains paramount. Delayed treatment is strongly associated with poor clinical outcomes (17). More importantly, the extension of the time window is not applicable to all patients but highly dependent on advanced neuroimaging screening (such as CTP, MRI-DWI) to confirm the presence of "ischemic penumbra" (i.e., salvageable brain tissue) (18). Many primary care hospitals lack these real-time imaging assessment capabilities, leading to delayed patient transfer or evaluation and missed treatment opportunities. As the predominant type of hemorrhagic stroke, the core of treatment strategies for cerebral hemorrhage lies in controlling bleeding, reducing intracranial pressure, preventing hematoma expansion, and managing complications, yet clinical efficacy remains a significant challenge. Current treatment approaches primarily include aggressive medical management and targeted surgical interventions, with all patients requiring multidisciplinary collaborative care in stroke units equipped with neurointensive care units (12). Medical treatment forms the foundation of cerebral hemorrhage management, with the primary goal being stabilization of vital signs. Key measures include emergency antihypertensive therapy to limit hematoma expansion, reversal of anticoagulant effects (such as using vitamin K or prothrombin complex for warfarin-related bleeding), and strict intracranial pressure management with complication prevention (19). Although aggressive medical management is the standard protocol, its effectiveness has significant limitations. Target values for antihypertensive therapy (e.g., rapidly reducing systolic blood pressure below 140mmHg) may lower hematoma expansion risk but have not been consistently shown to improve long-term neurological outcomes in all patients (20). For specific types of cerebral hemorrhage, surgical intervention serves as the primary approach to remove hematomas and relieve brain compression. Surgical options include craniotomy for hematoma evacuation and minimally invasive hematoma puncture drainage (typically combined with thrombolytic therapy to enhance drainage). The decision to operate is determined by critical factors such as hematoma size, location (e.g., cerebellar hemorrhage with brainstem compression or hydrocephalus often warrants surgery), neurological status, and age (21). However, surgical treatment faces significant challenges. The primary controversy lies in the difficulty of establishing definitive surgical indications and optimal timing. As demonstrated by the STICH series of studies, early surgical intervention offers uncertain benefits for most supratentorial hematomas (22).

2.3 Gut microbiota: A novel therapeutic approach for regulating central nervous system functions The gut microbiota refers to the complex microbial community colonizing the human gastrointestinal tract, with a cell count reaching 10^14-ten times the number of human cells. It encodes over 100 times more genes than the human genome, earning it the titles of "second brain" or "forgotten organ" (23). Primarily composed of bacteria, it also includes archaea, viruses, fungi, and protozoa (24). Its functions are remarkably diverse, ranging from nutrient metabolism (breaking down indigestible dietary fibers and producing beneficial substances like short-chain fatty acids) and vitamin synthesis (e.g., vitamin K and B vitamins) to immune system development, regulation, and defense against pathogens (25). Repairing and maintaining intestinal barrier function stands out as its most critical role. The complete intestinal barrier consists of four layers: mechanical (intestinal epithelial cells and tight junction proteins), chemical (mucus layer), immune (sIgA and lamina propria immune cells), and biological (the microbiota itself), effectively preventing harmful substances and pathogens from entering the bloodstream (26). The gut microbiota repairs the intestinal barrier through multiple mechanisms: its metabolic byproducts, particularly short-chain fatty acids (SCFAs) like butyric acid, serve as the primary energy source for colonic epithelial cells. These compounds promote cell proliferation and differentiation while directly enhancing the expression and assembly of tight junction proteins (e.g., Occludin, ZO-1), thereby reducing intestinal permeability (27). Furthermore, gut microbiota can thicken the chemical mucus layer by stimulating intestinal epithelial cells to secrete mucin (MUC2), while indirectly maintaining intestinal barrier integrity through immune regulation-such as promoting regulatory T cell (Treg) differentiation and reducing pro-inflammatory factor production.Disruption of gut microbiota is closely associated with impaired intestinal barrier function and serves as a key pathogenic mechanism for various diseases including inflammatory bowel disease (IBD), irritable bowel syndrome (IBS), metabolic syndrome, autoimmune disorders, and even neurological conditions (28).Microecological therapies based on gut microbiota theory aim to restore microbial balance for treating these conditions.Microbiotic preparations primarily include probiotics (live microorganisms like Bifidobacterium, Lactobacillus, and Clostridium butyricum), prebiotics (fructooligosaccharides, inulin), and synbiotics (combinations of probiotics and prebiotics) (29).These interventions work by directly supplementing beneficial bacteria, providing nutrients, or antagonizing pathogenic bacteria, representing first-line strategies for microbial regulation (30).A more effective approach is fecal microbiota transplantation (FMT), which involves transferring functional bacteria from healthy donors into the patient's gastrointestinal tract via enema, endoscopy, nasogastric tube, or capsule to reconstruct normal intestinal microecology (31).FMT is currently recognized as the most effective treatment for recurrent or refractory Clostridium difficile infections, with a cure rate exceeding 90% (32). Moreover, the clinical application of FMT in inflammatory bowel disease, metabolic syndrome, and other diseases is still in the exploratory stage, but its long-term safety, donor screening standardization, and mechanism of action require further research (33). Clostridium butyricum, a Gram-positive, spore-forming, obligate anaerobic bacillus, is named for its ability to produce large amounts of butyric acid and is one of the important strains in current probiotics (34). The core function of Clostridium butyricum is its colonization in the gut and production of large amounts of short-chain fatty acids, particularly butyric acid, which is a key substance for repairing intestinal barrier function (35). Its mechanisms of action include: 1.Direct enhancement of mechanical barrier: The butyric acid produced by Clostridium butyricum directly provides energy to colonic epithelial cells, promoting their proliferation and repair, and significantly upregulates the expression of tight junction proteins (such as ZO-1, Occludin), effectively reducing intestinal permeability and repairing "leaky gut" (36). 2.Regulation of immune response: Butyric acid has strong anti-inflammatory effects. It regulates gene expression by inhibiting histone deacetylase (HDAC) activity, promotes the differentiation and function of anti-inflammatory regulatory T cells (Treg), while suppressing pro-inflammatory signaling pathways such as NF-κB, reducing the production of pro-inflammatory factors like TNF-α and IL-6, thereby creating a favorable immune microenvironment for intestinal barrier repair (37). 3.Biological Antagonism: Clostridium butyricum competes with and suppresses pathogenic bacteria (e.g., Salmonella, Clostridium difficile) during colonization in the gut. The butyric acid it produces lowers intestinal pH, further inhibiting harmful bacteria and stabilizing the microbial community, thereby indirectly protecting the intestinal barrier (38). 4.Promoting Beneficial Bacteria Growth: Substances like butyric acid produced by Clostridium butyricum can also be utilized by other beneficial bacteria, promoting the growth and colonization of the entire beneficial microbial community to maintain intestinal microecological balance (38).

The gut-brain axis constitutes a complex bidirectional communication network connecting the central nervous system with the gut and its microbiota, centered on the integration of the microbiota-gut-brain axis concept (4). Its mechanisms primarily involve signal transmission through multiple pathways including neural (e.g., vagus nerve), endocrine (e.g., HPA axis and gut hormones), immune (e.g., cytokines), and microbial metabolic pathways (e.g., short-chain fatty acids (SCFAs) and neuroactive substances) (39). Dysregulation of the gut-brain axis has been demonstrated to be closely associated with various diseases, including irritable bowel syndrome (IBS) characterized by visceral hypersensitivity and motility abnormalities (40), inflammatory bowel disease (IBD) often accompanied by emotional comorbidities (41), autism spectrum disorder (ASD) with gastrointestinal symptoms and behavioral core symptoms (42), depression and anxiety related to microbiota dysbiosis and inflammation (43), and Parkinson's disease (PD) with pathological origins potentially originating in the gut (44). Recent studies support that gut microbiota interact with ischemic stroke through the gut-brain axis, thereby modulating stroke pathogenesis (45,46). Gut microbiota can influence host brain function and behavior through neural pathways (47), regulation of innate and adaptive immune responses (48), and their derived metabolites (49). Short-chain fatty acids (SCFAs) such as butyrate, as gut microbiota metabolites, alleviate neuroinflammation and brain injury by promoting regulatory T cell differentiation and secreting anti-inflammatory factors IL-10 and TGF-β, while suppressing pro-inflammatory Th1/Th17 responses and enhancing tight junction proteins Occludin and ZO-1 expression in the blood-brain barrier (45). Conversely, oxidized trimethylamine (TMAO), produced by gut microbiota through choline metabolism, activates the NLRP3 inflammasome to upregulate IL-1β and IL-18, thereby promoting atherosclerotic plaque formation and platelet aggregation, increasing ischemic stroke risk (50). Additionally, neuroactive substances like GABA produced by gut microbiota can regulate central nervous system inflammation via the vagus nerve (51). Compared to traditional stroke treatments, gut microbiota therapy for stroke breaks the time window limitation. Even days after stroke, restoring a youthful gut microbiome can reduce inflammation and promote recovery in stroke patients. This is largely mediated by bacterial metabolites, particularly SCFAs (52). Moreover, gut microbiota therapy for stroke can be achieved through easily accessible approaches like dietary modifications and probiotics, making it more accessible and scalable compared to traditional treatments constrained by equipment limitations (53). While existing studies have demonstrated the critical role of gut microbiota in stroke treatment (54), the mechanisms underlying its effects on improving physiological and behavioral functions in stroke patients remain insufficiently explored. A pressing question remains: How do gut microbiota and their metabolites specifically enhance stroke patient outcomes through neural pathways, immune system regulation, or other unexplored mechanisms?

Problem to be solved:

1. Key functional bacteria producing short-chain fatty acids play crucial roles in regulating gut microbiota, repairing intestinal barriers, and modulating immunity. Stroke disrupts intestinal motility, increases gut permeability, and activates resident immune cells, leading to microbial imbalance that transforms the gut microbiome into a more toxic state. Conversely, an ecologically disrupted gut microbiome communicates with the brain through the gut-brain axis (top-down signaling) to exacerbate stroke's harmful effects. However, the mechanisms by which gut functional bacteria improve stroke outcomes remain unclear. This study investigates the gut microbiota composition, intestinal barrier function, and inflammatory cytokine profiles in stroke patients and healthy individuals, aiming to elucidate the mechanisms of functional bacteria in stroke recovery and potentially provide new therapeutic approaches to overcome current treatment limitations.
2. The role of key functional bacteria producing short-chain fatty acids (SCFAs) in improving stroke prognosis: Poor post-stroke outcomes primarily involve motor and cognitive impairments caused by exacerbated neuroinflammation, as well as secondary infections resulting from gut microbiota metabolite translocation due to intestinal barrier damage (leaky gut) and systemic immune suppression. Through microbiota-targeted supplementation of SCFA-producing functional bacteria, we aim to reconstruct intestinal and host defense barriers. This research explores mechanisms including increased butyrate levels to inhibit microglial overactivation, promote regulatory T-cell differentiation, and enhance blood-brain barrier integrity, thereby improving stroke prognosis. The study identifies new therapeutic targets mediated by SCFAs and develops innovative neuroprotective strategies targeting the gut-brain axis.

Research objectives:

1. Utilize multi-omics technologies to elucidate post-stroke alterations in gut microbiota and host inflammatory responses from both host and microbial perspectives, and identify key functional bacteria and metabolites.
2. Investigate the regulatory effects of Clostridium butyricum on the gut microbiota and immune responses in stroke patients.
3. Investigate the mechanism by which Clostridium butyricum exerts neuroprotective effects through its metabolite short-chain fatty acids.
4. Investigate the modulating role of Clostridium butyricum in stroke patient prognosis.

2. Research Content, Research Approach, and Design research contents ：

1. To elucidate the patterns of post-stroke intestinal microbiota alterations and host inflammatory responses from both host and microbial perspectives, and to identify key functional bacteria and metabolites:

   Blood and stool samples were collected from stroke patients and healthy individuals, who were then categorized into a healthy control group and a stroke group based on laboratory test results. The study analyzed gut microbiota composition, fecal metabolomics, intestinal mucosal barrier function, and inflammatory cytokines to evaluate changes in gut microbiota and host inflammatory responses between groups, and to identify key functional bacteria and metabolites.
2. Clarifying the mechanism of key intestinal functional bacteria and fecal microbiota transplantation in improving the prognosis of stroke patients:

Establish a mouse model of stroke using key functional bacteria, key functional metabolites, and fecal microbiota transplantation (FMT) intervention. Analyze the intestinal microbiota composition, fecal metabolomics, intestinal mucosal barrier, and inflammatory cytokines in mice. Isolate brain and intestinal tissues to evaluate post-FMT recovery in both brain and gut, and identify the target sites of key functional metabolites after FMT.

Research ideas and design:

Proposed research plan:

1. Case selection:

Inclusion criteria: (1) First-time acute ischemic stroke patients with symptoms onset within 48 hours of hospital admission and initial sample collection; (2) Participants aged 18+ years old, regardless of gender; (3) Stroke patients with NIHSS scores ≥4; (4) Those who fully understand the study protocol and voluntarily participate.

Exclusion criteria: (1) Patients who took antibiotics or probiotics within one month prior to hospitalization or during follow-up; (2) Patients with infectious diseases such as pneumonia or urinary tract infections; (3) Patients who could not provide stool samples within three days after hospitalization or during three-month follow-up; (4) Patients with severe dysfunction of major organs including heart, lungs, liver, or kidneys; (5) Patients who did not provide or could not obtain informed consent; (6) Patients with a history of major gastrointestinal disorders; (7) Patients with severe neurological conditions; (8) Patients deemed unsuitable by investigators for participation in this clinical study.

Exclusion criteria: (1) Participants found to not meet inclusion criteria or meet exclusion criteria after enrollment; (2) Participants experiencing severe adverse events during the study must have the research paused.

ELIGIBILITY:
Inclusion Criteria:

(1) First-time acute ischemic stroke patients must have completed initial sample collection within 48 hours of symptom onset and hospital admission; (2) Participants must be aged 18 or older, with no gender restrictions; (3) Stroke patients must have a National Institutes of Health Stroke Scale (NIHSS) score of 4 or higher; (4) Participants must fully understand the study protocol and provide informed consent.

Exclusion Criteria:

(1) Patients who have taken antibiotics or probiotics within one month prior to hospitalization or during follow-up; (2) Patients with infectious diseases such as pneumonia or urinary tract infections; (3) Patients who cannot obtain stool samples within three days after hospitalization or during three-month follow-up; (4) Patients with severe dysfunction of major organs including heart, lungs, liver, or kidneys; (5) Patients who have not provided or are unable to provide informed consent; (6) Patients with a history of major gastrointestinal diseases; (7) Patients with other severe neurological disorders; (8) Patients deemed unsuitable by investigators to participate in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with ischemic stroke
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-11-19 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Gut microbiota composition | Within 48 hours of admission
  Fecal samples were processed using the QIAmp DNA Stool Fast Kit (QIAGEN, Hilden, Germany) for bacterial genome DNA extraction. The genomic library was constructed and sequenced on the MiSeq 300×2 V3 Kit (Illumina, USA) platform to comprehensively analyze the intestinal microbiota structure and composition. Bioinformatics analysis of the sequencing results included OTU generation and Rank-abundance analysis, sampling adequacy assessment, abundance and diversity analysis, microbial community differences, principal component analysis (PCA), hypothesis testing, and phylogenetic tree construction.

SECONDARY OUTCOMES:
Multiple cytokines | Within 48 hours of admission
  Using the Luminex 200 system with the Human27 Cytokine Combined Detection Kit, this method detects inflammatory factors, chemokines, and growth factors in host serum.

OTHER OUTCOMES:
Patient info | Before enrollment
  The patient's basic information includes age, sex, past history, present history, etc

CONTACTS AND LOCATIONS:
Overall Officials: Xiao MB Director of scientific research Department, Doctor, Principal Investigator — The Affiliated Hospital of Nantong University
Locations (1):
- Affiliated Hospital of Affiliated Hospital, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No